CLINICAL TRIAL: NCT03386981
Title: Study of the Metabolic Profile of Bone in Professional Athletes as a Function of the Kind of Physical Activity Performed
Brief Title: Metabolic Profile of Bone in Professional Athletes
Acronym: SportMarkers
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Elena Cittera, Scientific Direction, I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Other Study IDs: SportMarkers
Record Dates: First submitted 2017-12-05; First posted 2017-12-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Bone Disease, Metabolic; Physical Activity
Keywords: Energy metabolism; Homeostasis; Bone turnover markers
MeSH Terms: conditions — Bone Diseases, Metabolic; Motor Activity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and saliva will be collected under standard procedures as routine procedure independently decided by the team physicians. Waste material will be collected and analyzed for the aims of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Professional athletes: Professional athletes belonging to different discipline
  Interventions: Other: blood and saliva tests

INTERVENTIONS:
Other: blood and saliva tests — Blood and saliva will be tested for: bone turnover markers, cytokines, chemokines, adipokines, myokines and hormones regulating bone and energy metabolism

SUMMARY:
Physical activity is a key stimulus for bone metabolism through both direct mechanisms (e.g., as a result of the applied load and/or impact) and indirect mechanisms (e.g., the activation of several metabolic pathways and the production of several mediators and effectors that have systemic effects). However, different kinds of physical activity exert different effects on bone and endocrine system.

Aim of the study is to investigate the effects of different kinds of physical activity on bone metabolism and on the relationships existing between bone metabolism, energy metabolism, hormone profile, and organ functionality.

DETAILED DESCRIPTION:
Genetics explain about 70% of the inter-individual variance of bone mineral density (BMD) but maintenance and acquisition of bone mass strikingly depend on environmental factors as diet, calcium intake (in both quantitative and qualitative terms), and physical activity (PA). Among these, the biomechanical load generated by different kinds of PA represents the most important physiological stimulus able to increase bone mass and density.

Bone is a metabolically active tissue that undergoes to continuous remodeling throughout the coupling of resorption (operated by osteoclasts) and formation (operated by osteoblasts). Osteocytes, the quiescent form of osteoblasts, regulate the activity of the other two cell types and directly respond to load. Under normal conditions, resorption and formation are strikingly coupled and this guarantees an equilibrium between old bone matrix removal and new matrix deposition. This equilibrium is dependent upon several hormones and local mediators (e.g., cytokines, myokines, adipokines). Physiological (e.g., growth, aging, PA) and pathological conditions (e.g., metabolic diseases, bed rest, drugs) inbalance this equilibrium towards one side and, hence, affect bone mass. Regarding PA, for example, it is known that weight-bearing aerobic activity has positive effects on BMD and, hence, it is considered a preventive strategy against post-menopausal bone loss.

Differently from radiological imaging, that gives information about established architectural changes happened at a specific site in bone, biochemical and molecular markers of bone turnover give an instantaneous picture of the metabolic status of bone cells and, possibly, their immediate response to a stimulus.

Other than the bony response, PA activates several endocrine responses and particularly, the whole set of responses needed for managing the energy stores and to save the most nobile functions (e.g., brain, hearth). Hence, bone is subjected to the endocrine regulation of energy usage but, as recently discovered, being it the primary mechanosensor of load, it acts itself as an endocrine organ able to signal to other tissues and organs the changing environmental conditions.

Although several molecular aspects about the effects of PA on bone metabolism and the bone-energy cross-talk, a number of unresolved questions still exists. The study of different physiological models (i.e., athletes belonging to different disciplines) might allow the identification of common mechanisms regulating the response to PA and, from another side, to understand the physiological response to different stresses applied onto the muscle-skeletal apparatus.

The general aim of this study is to investigate the effects of different kinds of professional physical activity on bone metabolism and the relationship between bone metabolism, energy metabolism, hormone profile, and organ functionality.

The primary aim is to deepen the knowledge of the molecular mechanisms by which PA modulates bone metabolism. Specifically, this study will evaluate the bony effects of specific kinds of PA, over the time (over an entire season, over consecutive seasons, during different phases of a season), as well as the direct comparison of the bony effects of different kinds of PA and training.

Secondary aims are:

* to contextualize the modification of bone cell metabolism within the whole-body homeostatic profile. Particularly, markers of the energy metabolism and the inflammatory status (hormone, myokines, adipokines, cytokines, chemokines) will be evaluated.
* focused case-control studies will be conducted by including as little-active control the people belonging to the technical staff of the cooperating teams.

This is a perspective monocentric pilot study with different components:

* longitudinal perspective: repeated evaluations over the time
* case-control: comparison among different populations of athletes and technical staff Being based on already planned blood drawings (as independently decided by the team physicians), and since the researchers will use only waste material derived from these sample, the overall implant of the study is observational.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 yo
* healthy status
* caucasians

Exclusion Criteria:

* < 18 yo
* pregnancy status
* ongoing or previous (<5 years) neoplasia
* acute or chronic inflammatory pathologies
* primary metabolic diseases of bone
* recent bone fractures (< 6 months)
* chronic drugs
* recent drugs administration (< 2 months) for non steroidal anti-inflammatory drugs (NSAIDs) and steroids
* anxious-depressive conditions
* inability to understand the information given by the recruiting physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 subjects will be recruited. They will be recruited among professional athletes and technical staff of the cooperating teams
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02-04 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2027-02-04 (Estimated)

PRIMARY OUTCOMES:
Bone turnover markers | 0-36 Months
  different markers of bone turnover (osteocalcin, N-terminal type I pro-collagen, beta-crosslaps, osteopontin, bone-alkaline phosphatase, tartrate-resistant acid phosphatase 5b) will be tested depending on the group of subjects considered time-by-time

SECONDARY OUTCOMES:
myokines, adipokines, cytokines, chemokines, hormones regulating bone and energy metabolism | 0-36 Months
  different markers will be assayed depending on the group of subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Case Report Form (CRF) will be available

REFERENCES:
- [Background] Banfi G, Lombardi G, Colombini A, Lippi G. Bone metabolism markers in sports medicine. Sports Med. 2010 Aug 1;40(8):697-714. doi: 10.2165/11533090-000000000-00000. PMID 20632739
- [Background] Lombardi G, Lanteri P, Colombini A, Banfi G. Blood biochemical markers of bone turnover: pre-analytical and technical aspects of sample collection and handling. Clin Chem Lab Med. 2012 Feb 3;50(5):771-89. doi: 10.1515/cclm-2011-0614. PMID 22628324
- [Background] Chilibeck PD, Sale DG, Webber CE. Exercise and bone mineral density. Sports Med. 1995 Feb;19(2):103-22. doi: 10.2165/00007256-199519020-00003. PMID 7747001
- [Background] Murphy NM, Carroll P. The effect of physical activity and its interaction with nutrition on bone health. Proc Nutr Soc. 2003 Nov;62(4):829-38. doi: 10.1079/PNS2003304. PMID 15018482
- [Background] Snow CM, Williams DP, LaRiviere J, Fuchs RK, Robinson TL. Bone gains and losses follow seasonal training and detraining in gymnasts. Calcif Tissue Int. 2001 Jul;69(1):7-12. doi: 10.1007/s00223-001-0014-5. Epub 2001 Jun 5. PMID 11685427
- [Background] Shackelford LC, LeBlanc AD, Driscoll TB, Evans HJ, Rianon NJ, Smith SM, Spector E, Feeback DL, Lai D. Resistance exercise as a countermeasure to disuse-induced bone loss. J Appl Physiol (1985). 2004 Jul;97(1):119-29. doi: 10.1152/japplphysiol.00741.2003. PMID 15220316
- [Background] Lombardi G, Lanteri P, Graziani R, Colombini A, Banfi G, Corsetti R. Bone and energy metabolism parameters in professional cyclists during the Giro d'Italia 3-weeks stage race. PLoS One. 2012;7(7):e42077. doi: 10.1371/journal.pone.0042077. Epub 2012 Jul 27. PMID 22848709
- [Background] Seibel MJ. Biochemical markers of bone turnover: part I: biochemistry and variability. Clin Biochem Rev. 2005 Nov;26(4):97-122. PMID 16648882
- [Background] Corsetti R, Barassi A, Perego S, Sansoni V, Rossi A, Damele CA, Melzi D'Eril G, Banfi G, Lombardi G. Changes in urinary amino acids excretion in relationship with muscle activity markers over a professional cycling stage race: in search of fatigue markers. Amino Acids. 2016 Jan;48(1):183-92. doi: 10.1007/s00726-015-2077-z. Epub 2015 Aug 26. PMID 26306846
- [Background] Grasso D, Corsetti R, Lanteri P, Di Bernardo C, Colombini A, Graziani R, Banfi G, Lombardi G. Bone-muscle unit activity, salivary steroid hormones profile, and physical effort over a 3-week stage race. Scand J Med Sci Sports. 2015 Feb;25(1):70-80. doi: 10.1111/sms.12147. Epub 2013 Oct 31. PMID 24433517
- [Background] Lombardi G, Corsetti R, Lanteri P, Grasso D, Vianello E, Marazzi MG, Graziani R, Colombini A, Galliera E, Corsi Romanelli MM, Banfi G. Reciprocal regulation of calcium-/phosphate-regulating hormones in cyclists during the Giro d'Italia 3-week stage race. Scand J Med Sci Sports. 2014 Oct;24(5):779-87. doi: 10.1111/sms.12080. Epub 2013 May 7. PMID 23647316
- [Background] Lombardi G, Colombini A, Freschi M, Tavana R, Banfi G. Seasonal variation of bone turnover markers in top-level female skiers. Eur J Appl Physiol. 2011 Mar;111(3):433-40. doi: 10.1007/s00421-010-1664-7. Epub 2010 Sep 29. PMID 20878421
- [Background] Lombardi G, Lanteri P, Colombini A, Mariotti M, Banfi G. Sclerostin concentrations in athletes: role of load and gender. J Biol Regul Homeost Agents. 2012 Jan-Mar;26(1):157-63. PMID 22475109
- [Background] Lombardi G, Perego S, Luzi L, Banfi G. A four-season molecule: osteocalcin. Updates in its physiological roles. Endocrine. 2015 Mar;48(2):394-404. doi: 10.1007/s12020-014-0401-0. Epub 2014 Aug 27. PMID 25158976
- [Background] Walsh MC, Choi Y. Biology of the RANKL-RANK-OPG System in Immunity, Bone, and Beyond. Front Immunol. 2014 Oct 20;5:511. doi: 10.3389/fimmu.2014.00511. eCollection 2014. PMID 25368616
- [Background] Lombardi G, Sanchis-Gomar F, Perego S, Sansoni V, Banfi G. Implications of exercise-induced adipo-myokines in bone metabolism. Endocrine. 2016 Nov;54(2):284-305. doi: 10.1007/s12020-015-0834-0. Epub 2015 Dec 30. PMID 26718191
- [Background] Fang S, Deng Y, Gu P, Fan X. MicroRNAs regulate bone development and regeneration. Int J Mol Sci. 2015 Apr 13;16(4):8227-53. doi: 10.3390/ijms16048227. PMID 25872144
- [Background] Allison RJ, Farooq A, Hamilton B, Close GL, Wilson MG. No association between vitamin D deficiency and markers of bone health in athletes. Med Sci Sports Exerc. 2015 Apr;47(4):782-8. doi: 10.1249/MSS.0000000000000457. PMID 25058327